CLINICAL TRIAL: NCT01127230
Title: Comparison Between Celution Preparation and Manual Preparation of Adipocyte Derived Regenerative Cells, Using Stromal Vascular Fraction Cell Counts (COMPARE)
Acronym: COMPARE
Status: Completed | Type: Observational
Sponsor: Novena Medical Center (Network)
Responsible Party: Dr Tan Kok Leong, Life Source Medical Centre
Other Study IDs: 01-2010/03/14-S0001
Record Dates: First submitted 2010-05-19; First posted 2010-05-20 (Estimated); Last update posted 2010-07-19 (Estimated); Status verified 2010-07

CONDITIONS: Obesity
Keywords: ADRC; adipocyte derived regenerative cells; stem cells; liposuction; Cytori; Celution; Lipoaspirate is obtained from patients who have opted for liposuction and consent to donate the lipoasirate for this study, which would otherwise be discarded.
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Biospecimen Retention: Samples With DNA — Lipoaspirate from liposuction.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Liposuction patients: Patients who already opted and are scheduled for liposuction.

SUMMARY:
This scientific study is meant to establish correlation in Stromal Vascular Fraction (SVF) cell counts between our manual method of harvesting and Cytori's Celution automated system.

Future scientific studies involving Adipocyte Derived Regenerative Cells (ADRCs) will be based on SVF cell counts from the more economical manual method of harvesting if this study shows good correlation.

DETAILED DESCRIPTION:
This study requires lipoaspirate obtained from liposuction. Lipoaspirate is typically discarded in the biohazard waste disposal system. We will be using the lipoaspirate (which would otherwise be discarded) in this study.

Lipoaspirate contains adipose tissues. With a suitable enzymatic separation method, stromal vascular fraction (SVF) can be separated from the adipose cells (adipocyte).

Adipocyte derived regenerative cells has been isolated from the stromal vascular fraction (SVF) of adipose tissues. There are two methods of obtaining the SVF from the adipose tissue in this study. One is called the manual preparation and the other the Celution preparation. The Celution preparation is an automated system, providing a constant standard by which to compare the manual preparation of SVF. This study aims to establish correlation between the manual preparation and Celution preparation.

The purpose of establishing correlation is to allow the manual preparation of SVF to be used in future scientific studies. The manual preparation has the advantage of being more economical than the Celution automated system.

In future scientific studies, we hope to establish correlation between survival rates of fat graft and SVF cell counts. Currently fat grafting is an accepted List A aesthetic procedure in Singapore to enhance facial features and in breast augmentation. However results vary widely among patients, and seems unpredictable. A possible hypothesis is that the survivability of the fat graft is dependent on the number of naturally occurring ADRCs found in the fat graft. In the future we hope to conduct a scientific study on this hypothesis using the manual preparation.

The secondary purpose for this study is to correlate SVF cell counts with the age, sex, weight, BMI and anatomical area of liposuction.

ELIGIBILITY:
Inclusion Criteria:

* patients who already opted for liposuction
* patients who consents to donate the lipoaspirate after liposuction
* patients more than 21 years of age

Exclusion Criteria:

* patients with history of organ failure
* patients with history of carcinoma
* patients who are pregnant

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Liposuction Patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Stromal Vascular Fraction Cell Count Ratio | 1 day
  SVF cell count Ratio = SVF cell count from Cytori's Celution : SVF cell count from manual preparation

SECONDARY OUTCOMES:
Stromal Vascular Fraction Cell Count Age Comparison . | 1 day
  SVF cell counts differences in different age groups

CONTACTS AND LOCATIONS:
Overall Officials: Kok Leong Tan, MBBS, Principal Investigator — Life Source Medical Centre
Locations (1):
- Life Source Medical Centre, Singapore, Singapore, Singapore